CLINICAL TRIAL: NCT01108146
Title: Monocentric, Double-blind Placebo-Controlled, Randomized Cross-Sectional Clinical Trial of Hydrocortisone (10 and 30 mg/d) in Outpatients With Posttraumatic-Stress-Disorder (PTSD)
Brief Title: Hydrocortisone in the Treatment of Intrusions in Patients With Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Christian Schmahl, Prof. Dr., Central Institute of Mental Health, Mannheim
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HPA-PTSD-1
Record Dates: First submitted 2010-02-16; First posted 2010-04-21 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Drug: Hydrocortisone 10 mg
  Group 1: Administration of Hydrocortisone and/or Placebo in the following order:
  1 week placebo-1 week hydrocortisone 10 mg/d -1 week placebo - 1 week hydrocortisone 30 mg/d
  Interventions: Drug: Arm 1 Hydrocortisone 10 mg
- Arm 2 (Experimental): Drug: Hydrocortisone 30 mg
  Group 2: Administration of Hydrocortisone and/or Placebo in the following order:
  1 week hydrocortisone 30 mg/d- 1 week placebo - 1 week hydrocortisone 10 mg/d - 1 week placebo
  Interventions: Drug: Arm 2 Hydrocortisone 30 mg

INTERVENTIONS:
Drug: Arm 1 Hydrocortisone 10 mg — Group 1: Administration of Hydrocortisone and/or Placebo in the following order:
  1 week placebo- 1 week 10 mg hydrocortisone - 1 week placebo - 1 week 30 mg hydrocortisone
  Arms: Arm 1
Drug: Arm 2 Hydrocortisone 30 mg — Drug: Hydrocortisone 30 mg
  Group 2: Administration of Hydrocortisone and/or Placebo in the following order:
  1 week hydrocortisone 30 mg/d- 1 week placebo - 1 week hydrocortisone 10 mg/d - 1 week placebo
  Arms: Arm 2

SUMMARY:
To test overall efficacy of hydrocortisone on reexperience of traumatic memories (intrusions) and overall symptomatology in patients meeting criteria of complex chronic PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent
* Female patients with PTSD according to DSM-IV criteria (see Appendix 2).
* 18-45 years
* Intrusions (according to IES-R subscale Intrusions: Value: > 7
* Ability of subject to understand character and individual consequences of the clinical trial
* No participation in another clinical trial (up from 30 days before this trial)

Exclusion Criteria:

* Lifetime diagnosis schizophrenia according to DSM-IV
* Mental retardation
* Body mass index < 16.5
* Current drug and alcohol abuse and addiction
* Life-threatening self-injurious behavior in the last 4 months
* Suicide attempt with the strong intention to die in the last 4 months.
* Following diseases in anamnesis: stomach ulcera or intestinal ulcera, pancreatitis, corticoid-induced psychosis, severe osteoporosis, severe hyper-tension, heart failure, myasthenia gravis, asthma bronchiale, glaucoma, cataract, diabetes mellitus, herpes simples, herpes zoster (viremic phase), renal transplantation.
* Any pretreatment with hydrocortisone in the last 4 weeks prior to the first administration of Investiga-tional Medicinal Product.
* Following current medication: cardiac glycosides, saluretics, antidiabetics, cumarin-derivatives, rifampicine, phenytoine, barbiturates, primidone, NSAID, salicylate and indometacine, atropine, praziquantel, chloroquine, hydroxychloroquine, mefloquine, somatropine, protireline, cyclosporine, non-depolarising muscle relaxants.
* Pregnancy or lactation period
* Inadequate birth control (Adequate birth control: implants, injectables, combined oral contraceptives, intrauterine devices (IUDs), sexual abstinence or vasectomised partner)
* Shift working
* Intercontinental travel within 2 weeks prior to enrollment (to avoid jet-lag)
* History of hypersensitivity to investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.
* No subject will be allowed to enrol in this trial more than once.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Reduction of the frequency and intensity of intrusions assessed with the subscale Intrusions of the Impact of Event Scale (IES-R) | 4 Years

SECONDARY OUTCOMES:
Reduction of the overall PTSD symptomatology assessed with the IES-R and the Posttraumatic Diagnostic Scale (PDS) | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Schmahl, MD, Principal Investigator — Central Insitute of Mental Health, Dpt. of Psychosomatic and Psychotherapeutic Medicine
Locations (1):
- Central Institute of Mental Health, Dpt. of Psychosomatic and Psychotherapeutic Medicine, Mannheim, Germany

REFERENCES:
- [Derived] Ludascher P, Schmahl C, Feldmann RE Jr, Kleindienst N, Schneider M, Bohus M. No evidence for differential dose effects of hydrocortisone on intrusive memories in female patients with complex post-traumatic stress disorder--a randomized, double-blind, placebo-controlled, crossover study. J Psychopharmacol. 2015 Oct;29(10):1077-84. doi: 10.1177/0269881115592339. Epub 2015 Jul 6. PMID 26152322